CLINICAL TRIAL: NCT07208682
Title: Does Retropubic Hydrodissection Decrease Trocar-induced Bladder Perforation Rates During Placement of Retropubic Midurethral Slings? A Randomized Controlled Trial
Brief Title: Retropubic Hydrodissection and Trocar-induced Bladder Perforation During Retropubic Midurethral Slings
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Emily Wu, Physician, University of Massachusetts, Worcester
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: STUDY00002369
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Bladder Perforation; Retropubic Midurethral Sling; Retropubic Hydrodissection
Keywords: bladder perforation; retropubic midurethral sling; retropubic hydrodissection

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Retropubic hydrodissection (Active Comparator): subjects would receive a total of 60cc sterile injectable saline in the retropubic space using a 20g spinal needle placed in the anticipated path of the trocars
  Interventions: Procedure: retropubic hydrodissection
- No retropubic hydrodissection (No Intervention): this group would not receive retropubic hydrodissection

INTERVENTIONS:
Procedure: retropubic hydrodissection — subjects would receive retropubic hydrodissection prior to passage of the trocars. A total of 60cc of sterile injectable saline would be injected in the retropubic space with a 20g spinal needle along the anticipated path of the trocar.
  Arms: Retropubic hydrodissection

SUMMARY:
Retropubic midurethral slings are a common and effective treatment for stress urine incontinence. The trocar that is attached to the mesh material can hit the bladder which is called a perforation. While there are no known long-term adverse outcomes from trocar-induced bladder perforations, it can prolong operative time and bleeding. At academic institutions, it has been reported that trocar-induced perforations occurs in the range of 14-34% of the time. This study is a randomized controlled trial to see if an intervention can decrease trocar-induced bladder perforation rates. The primary outcome of this study is to measure trocar-induced bladder perforations in subjects undergoing a retropubic midurethral sling. Subjects would be randomized to either receive the hydrodissection in a standardized manner or to not receive it. Secondary outcomes include bothersome urinary symptoms, pain, estimated blood loss during surgery, and voiding trial results

DETAILED DESCRIPTION:
All female adult subjects presenting to the UMass urogynecology clinic for scheduled retropubic midurethral sling surgery will be eligible for recruitment. Subjects will also be recruited if they are fluent in English and/or Spanish, and able to fill out consent and questionnaires. Subjects would be excluded if they are limited English or Spanish proficiency to participate in the study, pregnant, or having concurrent surgery for malignancy.

At the time of enrollment which would be done at a preoperative visit, subjects would be asked to fill out a baseline urinary symptom questionnaire (UDI-6). On the day of surgery, each subject would be randomized via computer-generated randomization table to either the intervention group (receiving retropubic hydrodissection) or no intervention group.

The method of hydrodissection is described as the following: After the peri-urethral dissection is performed and the bladder is continuously drained and emptied via Foley catheter, a 20-gauge spinal needle is used to administer a total of 60ml of sterile injectable saline in the retropubic space. The surgeon will insert the needle approximately 2-3cm on each side of the midline just above the pubic symphysis. With another hand in the vagina, the surgeon will guide the needle to the retropubic space and infiltrate along the anticipated path of the trocar and inject 30ml of saline in the retropubic space on each side.

Intraoperative data collected includes number of trocar-induced bladder

ELIGIBILITY:
Inclusion Criteria:

* scheduled for retropubic midurethral sling

Exclusion Criteria:

* cognitive or intellectual impairment that would hinder ability to complete questionnaires or be consented
* having concurrent surgery for malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — female
Enrollment: 300 (Estimated)
Dates: Start 2025-04-03 (Actual); Primary Completion 2027-04 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
trocar-induced bladder perforation | during the surgery
  the number of trocar-induced bladder perforations during one case would be measured

CONTACTS AND LOCATIONS:
Locations (1):
- University of Massachusetts Memorial Medical Center, Worcester, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No